CLINICAL TRIAL: NCT00195702
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Human Anti-TNF Monoclonal Antibody Adalimumab in Rheumatoid Arthritis Patients Currently Receiving Treatment With Methotrexate
Brief Title: Efficacy and Safety of Adalimumab in Patients With Active Rheumatoid Arthritis Treated Concomitantly With Methotrexate.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DE019
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2010-03-01 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- DB adalimumab 20 mg ew (Experimental): Subjects received 20 mg adalimumab subcutaneously (SC) once weekly (ew) and concomitant methotrexate (MTX) during the double-blind (DB) phase.
  Interventions: Biological: Adalimumab
- DB adalimumab 40 mg eow (Experimental): Subjects received 40 mg adalimumab subcutaneously (SC) every other week (eow) and concomitant methotrexate (MTX) during the double-blind (DB) phase. Subjects received placebo injections SC and concomitant MTX on the alternate weeks during the DB phase.
  Interventions: Biological: Adalimumab
- DB placebo ew (Placebo Comparator): Subjects received placebo subcutaneously (SC) once weekly (ew) and concomitant methotrexate (MTX) during the double-blind (DB) phase.
  Interventions: Drug: Placebo
- DB adalimumab 20 mg ew/OL adalimumab 40 mg eow (Experimental): Subjects received adalimumab 20 mg subcutaneously (SC) once weekly (ew) during the double-blind (DB) phase, then adalimumab 40 mg SC every other week (eow) during the open-label (OL) extension phase, along with concomitant methotrexate (MTX).
  Interventions: Biological: Adalimumab
- DB adalimumab 40 mg eow/OL adalimumab 40 mg eow (Experimental): Subjects received adalimumab 40 mg subcutaneously (SC) every other week (eow) with placebo on alternate weeks during the double-blind (DB) phase, then adalimumab 40 mg SC eow during the open-label (OL) extension phase, along with concomitant methotrexate (MTX).
  Interventions: Biological: Adalimumab
- DB placebo ew/OL adalimumab 40 mg eow (Experimental): Subjects received placebo subcutaneously (SC) once weekly (ew) during the double-blind phase, then adalimumab 40 mg SC every other week (eow) during the open-label (OL) extension phase, along with concomitant methotrexate (MTX).
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab — Self-administered, subcutaneous injection of 20 mg adalimumab (1.6 mL/injection) once weekly (ew) for up to 52 weeks.
  Other Names: ABT-D2E7; Humira
  Arms: DB adalimumab 20 mg ew
Biological: Adalimumab — Self-administered, subcutaneous injection of 40 mg adalimumab (1.6 mL/injection) every other week (eow) for up to 52 weeks.
  Other Names: ABT-D2E7; Humira
  Arms: DB adalimumab 40 mg eow
Drug: Placebo — Self-administered, subcutaneous injection of placebo (1.6 mL/injection) once weekly (ew) for up to 52 weeks.
  Arms: DB placebo ew
Biological: Adalimumab — Self-administration, subcutaneous (SC) injection of adalimumab 20 mg (1.6 mL/injection) once weekly (ew) for 52 weeks, followed by self-administration, SC injection of adalimumab 40 mg (0.8 mL/injection) every other week (eow) for up to Week 520.
  Other Names: ABT-D2E7; Humira
  Arms: DB adalimumab 20 mg ew/OL adalimumab 40 mg eow
Biological: Adalimumab — Self-administration, subcutaneous (SC) injection of adalimumab 40 mg (1.6 mL/injection) every other week (eow) (with a placebo 1.6 mL/injection on alternate weeks) for 52 weeks, followed by self-administration, SC injection of adalimumab 40 mg (0.8 mL injection) eow for up to Week 520.
  Other Names: ABT-D2E7; Humira
  Arms: DB adalimumab 40 mg eow/OL adalimumab 40 mg eow
Biological: Adalimumab — Self-administration, subcutaneous (SC) injection of placebo solution (1.6 mL/injection) once weekly (ew) for 52 weeks, followed by self-administration, SC injection of adalimumab 40 mg (0.8 mL/injection) every other week (eow) for up to Week 520.
  Other Names: ABT-D2E7; Humira
  Arms: DB placebo ew/OL adalimumab 40 mg eow

SUMMARY:
The purpose of the study was to assess the safety, immunogenicity, and clinical efficacy of adalimumab compared with placebo (during double-blind phase) and to to evaluate the long-term safety and maintenance of efficacy following repeated administration of adalimumab (during open-label extension phase) in patients with persistently active rheumatoid arthritis who were receiving concurrent methotrexate therapy.

DETAILED DESCRIPTION:
This was a 10-year study which had an initial 52-week, double-blind, placebo-controlled phase followed by an open-label extension phase up to 9 years in duration. Data were analyzed for the double-blind phase using all patients who were randomized and received at least one dose of study drug through Week 52 and for all patients who received at least one dose of adalimumab during the 10-year study (the Intent-to-Treat [ITT] population).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older and in good health (Investigator discretion) with a recent stable medical history
* Met American College of Rheumatology (ACR) criteria for diagnosis of active rheumatoid arthritis (RA) and had at both screening and baseline visits >=6 swollen joints and >=9 tender joints, despite a minimum of 3-months treatment with methotrexate (MTX). (Distal interphalangeal joints [DIPs] were not to be included in joint count for inclusion. The screening and baseline visits could be 3 to 28 days apart for patients not previously receiving disease-modifying anti-rheumatic drugs [DMARDs] other than MTX or 4 to 6 weeks for patients requiring a DMARD washout period.)
* Insufficient efficacy with MTX 12.5 to 25 mg per week (10 mg per week if MTX intolerant).
* If patient on a second-line treatment (DMARD) other than MTX, he/she had to discontinue it for at least 28 days before the baseline visit (the washout period).
* Treatment with oral folic acid 1-3 mg/day or, if appropriate, up to 10 mg leucovorin per week.
* Both rheumatoid factor positivity and a C-reactive protein value >=1 mg/dL, or at least one joint erosion on X-ray.

Exclusion Criteria:

* Subject considered by the investigator, for any reason, to be an unsuitable candidate for the study.
* Female subject who was pregnant or breast-feeding or considering becoming pregnant.
* Preceding treatment with any tumor necrosis factor (TNF) antagonist, including adalimumab.
* Prior exposure to alkylating agents, such as chlorambucil or cyclophosphamide.
* Intra-articular, intramuscular, or intravenous administration of corticosteroids within 4 weeks prior to the screening visit.
* Subject was wheelchair bound or bedridden.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 619 (Actual)
Dates: Start 2000-02; Primary Completion 2002-09 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Redden, MD, PhD, Study Director — Abbott
Locations (87):
- United States (76):
  - Site Ref # / Investigator 424, Huntsville, Alabama
  - Site Ref # / Investigator 2510, Mobile, Alabama
  - Site Ref # / Investigator 60729, Phoenix, Arizona
  - Site Ref # / Investigator 725, Scottsdale, Arizona
  - Site Ref # / Investigator 60736, Anaheim, California
  - Site Ref # / Investigator 360, Escondido, California
  - Site Ref # / Investigator 714, La Jolla, California
  - Site Ref # / Investigator 469, La Jolla, California
  - Site Ref # / Investigator 419, Palm Desert, California
  - Site Ref # / Investigator 492, San Jose, California
  - Site Ref # / Investigator 60734, San Louis Obispo, California
  - Site Ref # / Investigator 60739, Van Nuys, California
  - Site Ref # / Investigator 712, Danbury, Connecticut
  - Site Ref # / Investigator 710, Aventura, Florida
  - Site Ref # / Investigator 498, Dunedin, Florida
  - Site Ref # / Investigator 499, Orlando, Florida
  - Site Ref # / Investigator 729, Tampa, Florida
  - Site Ref # / Investigator 463, Zephyrhills, Florida
  - Site Ref # / Investigator 2436, Boise, Idaho
  - Site Ref # / Investigator 485, Idaho Falls, Idaho
  - Site Ref # / Investigator 60732, Chicago, Illinois
  - Site Ref # / Investigator 726, Springfield, Illinois
  - Site Ref # / Investigator 2506, Indianapolis, Indiana
  - Site Ref # / Investigator 732, South Bend, Indiana
  - Site Ref # / Investigator 60730, Shawnee Mission, Kansas
  - Site Ref # / Investigator 467, Wichita, Kansas
  - Site Ref # / Investigator 494, Wichita, Kansas
  - Site Ref # / Investigator 491, Lexington, Kentucky
  - Site Ref # / Investigator 2508, Portland, Maine
  - Site Ref # / Investigator 392, Baltimore, Maryland
  - Site Ref # / Investigator 354, Cumberland, Maryland
  - Site Ref # / Investigator 730, Wheaton, Maryland
  - Site Ref # / Investigator 465, Burlington, Massachusetts
  - Site Ref # / Investigator 2512, Worcester, Massachusetts
  - Site Ref # / Investigator 471, Grand Rapids, Michigan
  - Site Ref # / Investigator 473, Kalamazoo, Michigan
  - Site Ref # / Investigator 731, Kansas City, Missouri
  - Site Ref # / Investigator 502, St Louis, Missouri
  - Site Ref # / Investigator 482, St Louis, Missouri
  - Site Ref # / Investigator 371, St Louis, Missouri
  - Site Ref # / Investigator 487, Omaha, Nebraska
  - Site Ref # / Investigator 353, Concord, New Hampshire
  - Site Ref # / Investigator 364, Dover, New Hampshire
  - Site Ref # / Investigator 60726, Mercerville, New Jersey
  - Site Ref # / Investigator 358, Voorhees Township, New Jersey
  - Site Ref # / Investigator 483, Rochester, New York
  - Site Ref # / Investigator 512, Durham, North Carolina
  - Site Ref # / Investigator 340, Greensboro, North Carolina
  - Site Ref # / Investigator 461, Raleigh, North Carolina
  - Site Ref # / Investigator 500, Raleigh, North Carolina
  - Site Ref # / Investigator 60731, Raleigh, North Carolina
  - Site Ref # / Investigator 60737, Salisbury, North Carolina
  - Site Ref # / Investigator 456, Mayfield Village, Ohio
  - Site Ref # / Investigator 470, Oklahoma City, Oklahoma
  - Site Ref # / Investigator 60723, Oklahoma City, Oklahoma
  - Site Ref # / Investigator 422, Eugene, Oregon
  - Site Ref # / Investigator 60735, Colmar, Pennsylvania
  - Site Ref # / Investigator 2507, Duncansville, Pennsylvania
  - Site Ref # / Investigator 717, East Norriton, Pennsylvania
  - Site Ref # / Investigator 352, Mechanicsburg, Pennsylvania
  - Site Ref # / Investigator 480, Wexford, Pennsylvania
  - Site Ref # / Investigator 2511, Wyomissing, Pennsylvania
  - Site Ref # / Investigator 60724, Wyomissing, Pennsylvania
  - Site Ref # / Investigator 718, Charleston, South Carolina
  - Site Ref # / Investigator 460, Memphis, Tennessee
  - Site Ref # / Investigator 462, Nashville, Tennessee
  - Site Ref # / Investigator 716, Austin, Texas
  - Site Ref # / Investigator 60728, Galveston, Texas
  - Site Ref # / Investigator 2509, Houston, Texas
  - Site Ref # / Investigator 510, Houston, Texas
  - Site Ref # / Investigator 60725, Falls Church, Virginia
  - Site Ref # / Investigator 711, Richmond, Virginia
  - Site Ref # / Investigator 509, Seattle, Washington
  - Site Ref # / Investigator 356, Spokane, Washington
  - Site Ref # / Investigator 464, Tacoma, Washington
  - Site Ref # / Investigator 60738, Kenosha, Wisconsin
- Canada (11):
  - Site Ref # / Investigator 475, Calgary, Alberta
  - Site Ref # / Investigator 495, Penticton, British Columbia
  - Site Ref # / Investigator 2496, Richmond, British Columbia
  - Site Ref # / Investigator 2495, Winnipeg, Manitoba
  - Site Ref # / Investigator 496, Halifax, Nova Scotia
  - Site Ref # / Investigator 444, Newmarket, Ontario
  - Site Ref # / Investigator 2497, Toronto, Ontario
  - Site Ref # / Investigator 478, Toronto, Ontario
  - Site Ref # / Investigator 421, Toronto, Ontario
  - Site Ref # / Investigator 363, Montreal, Quebec
  - Site Ref # / Investigator 60702, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Smolen J, Fleischmann R, Aletaha D, Li Y, Zhou Y, Sainsbury I, Galindo IL. Disease activity improvements with optimal discriminatory ability between treatment arms: applicability in early and established rheumatoid arthritis clinical trials. Arthritis Res Ther. 2019 Nov 10;21(1):231. doi: 10.1186/s13075-019-2005-9. PMID 31707982
- [Derived] Keystone EC, Breedveld FC, van der Heijde D, van Vollenhoven RF, Emery P, Smolen JS, Sainsbury I, Florentinus S, Kupper H, Chen K, Kavanaugh A. Achieving comprehensive disease control in patients with early and established rheumatoid arthritis treated with adalimumab plus methotrexate versus methotrexate alone. RMD Open. 2017 Sep 26;3(2):e000445. doi: 10.1136/rmdopen-2017-000445. eCollection 2017. PMID 29018564
- [Derived] Burmester GR, Landewe R, Genovese MC, Friedman AW, Pfeifer ND, Varothai NA, Lacerda AP. Adalimumab long-term safety: infections, vaccination response and pregnancy outcomes in patients with rheumatoid arthritis. Ann Rheum Dis. 2017 Feb;76(2):414-417. doi: 10.1136/annrheumdis-2016-209322. Epub 2016 Jun 23. PMID 27338778
- [Derived] Emery P, Kavanaugh A, Bao Y, Ganguli A, Mulani P. Comprehensive disease control (CDC): what does achieving CDC mean for patients with rheumatoid arthritis? Ann Rheum Dis. 2015 Dec;74(12):2165-74. doi: 10.1136/annrheumdis-2014-205302. Epub 2014 Aug 19. PMID 25139667
- [Derived] Landewe R, Ostergaard M, Keystone EC, Florentinus S, Liu S, van der Heijde D. Analysis of integrated radiographic data from two long-term, open-label extension studies of adalimumab for the treatment of rheumatoid arthritis. Arthritis Care Res (Hoboken). 2015 Feb;67(2):180-6. doi: 10.1002/acr.22426. PMID 25073879
- [Derived] Keystone EC, van der Heijde D, Kavanaugh A, Kupper H, Liu S, Guerette B, Mozaffarian N. Clinical, functional, and radiographic benefits of longterm adalimumab plus methotrexate: final 10-year data in longstanding rheumatoid arthritis. J Rheumatol. 2013 Sep;40(9):1487-97. doi: 10.3899/jrheum.120964. Epub 2013 Jul 1. PMID 23818718
- [Derived] Keystone EC, Kavanaugh A, Weinblatt ME, Patra K, Pangan AL. Clinical consequences of delayed addition of adalimumab to methotrexate therapy over 5 years in patients with rheumatoid arthritis. J Rheumatol. 2011 May;38(5):855-62. doi: 10.3899/jrheum.100752. Epub 2011 Feb 1. PMID 21285171

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 95 sites in the United States and Canada between February 2000 and August 2001.
Pre-assignment Details: Eligible subjects who were taking disease-modifying anti-rheumatic drugs (DMARDs) other than methotrexate (MTX) entered a 4- to 6-week washout period, during which previous DMARDs (except MTX) were discontinued. Subjects who were not taking DMARDs, other than MTX, entered directly into the 52-week double-blind treatment period of the study.
Groups:
- DB Adalimumab 20 mg ew: Subjects received adalimumab 20 mg every week (ew) and concomitant methotrexate (MTX) during the 52-week double-blind phase.
- DB Adalimumab 40 mg Eow: Subjects received adalimumab 40 mg every other week (eow) and concomitant methotrexate (MTX) during the 52-week double-blind phase.
- DB Placebo ew: Subjects received placebo every week and concomitant methotrexate (MTX) during the 52-week double-blind phase.
- DB Adalimumab 20 mg ew/OL Adalimumab 40 mg Eow: Subjects received adalimumab 20 mg weekly (ew) during the double-blind (DB) phase, then received adalimumab 40 mg every other week (eow) during the open-label (OL) extension phase. Subjects received concomitant methotrexate (MTX) during both phases of the study.
- DB Adalimumab 40 mg Eow/OL Adalimumab 40 mg Eow: Subjects received adalimumab 40 mg every other week (eow) during the double-blind (DB) phase, then received adalimumab 40 mg every other week (eow) during the open-label (OL) extension phase. Subjects received concomitant methotrexate (MTX) during both phases of the study.
- DB Placebo ew/OL Adalimumab 40 mg Eow: Subjects received placebo weekly (ew) during the double-blind (DB) phase, then received adalimumab 40 mg every other week (eow) during the open-label (OL) extension phase. Subjects received concomitant methotrexate (MTX) during both phases of the study.
Period: Double-blind Phase
Arm/Group | DB Adalimumab 20 mg ew | DB Adalimumab 40 mg Eow | DB Placebo ew | DB Adalimumab 20 mg ew/OL Adalimumab 40 mg Eow | DB Adalimumab 40 mg Eow/OL Adalimumab 40 mg Eow | DB Placebo ew/OL Adalimumab 40 mg Eow
Started | 212 (For all groups, started indicates when the subjects entered the 52-week double-blind phase.) | 207 | 200 | 0 | 0 | 0
Completed | 168 | 159 | 140 | 0 | 0 | 0
Not Completed | 44 | 48 | 60 | 0 | 0 | 0
Period: Open-label Extension Phase
Arm/Group | DB Adalimumab 20 mg ew | DB Adalimumab 40 mg Eow | DB Placebo ew | DB Adalimumab 20 mg ew/OL Adalimumab 40 mg Eow | DB Adalimumab 40 mg Eow/OL Adalimumab 40 mg Eow | DB Placebo ew/OL Adalimumab 40 mg Eow
Started | 0 | 0 | 0 | 165 (3 subjects completed the double-blind phase but did not enter the open-label extension phase.) | 158 (1 subject completed the double-blind phase but did not enter the open-label extension phase.) | 134 (6 subjects completed the double-blind phase but did not enter the open-label extension phase.)
Completed | 0 | 0 | 0 | 66 | 80 | 56
Not Completed | 0 | 0 | 0 | 99 | 78 | 78

BASELINE CHARACTERISTICS:
Groups:
- DB Adalimumab 20 mg ew: Subjects received adalimumab 20 mg every week (ew) and concomitant methotrexate (MTX) during the 52-week double-blind treatment phase.
- Total: Total of all reporting groups
Arm/Group | DB Adalimumab 20 mg ew | DB Adalimumab 40 mg Eow | DB Placebo ew | Total
Number analyzed (Participants) | 212 | 207 | 200 | 619
Age, Customized [Number; unit: participants]
  < 40 years | 10 | 27 | 18 | 55
  Between 40 and 64 years | 150 | 115 | 137 | 402
  Between 65 and 74 years | 41 | 54 | 35 | 130
  >= 75 years | 11 | 11 | 10 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 158 | 146 | 464
  Male | 52 | 49 | 54 | 155

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Meeting American College of Rheumatology 20% (ACR20) Response Criteria at Week 24
Description: Patients were responders if they had: >= 20% improvement in tender joint count; >= 20% improvement in swollen joint count; and >= 20% improvement in at least 3 of 5 remaining ACR core measures: patient assessment of pain; patient global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and acute phase reactant: C-reactive protein. Patients withdrawing early or receiving additional disease-modifying anti-rheumatic drugs (DMARDs) after Week 16 were non-responders.
Time Frame: Week 24
Population: Full analysis set, defined as all subjects who were randomized and received at least one injection of study drug. Observed data were analyzed.
Measure: Number; unit: Participants
Arm/Group | DB Adalimumab 20 mg ew | DB Adalimumab 40 mg Eow | DB Placebo ew
Number analyzed (Participants) | 212 | 207 | 200
Participants | 129 | 131 | 59
Statistical Analysis 1: Comparison: DB Adalimumab 20 mg ew vs DB Placebo ew; The 3 primary efficacy variables were considered in a hierarchical order, with the ACR20 response tested first. The ACR20 response rate at Week 24 was initially assessed using Pearson's chi-squared test at a significance level of 0.05. If significant, pairwise comparisons between each adalimumab dose group and the placebo group were performed; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: DB Adalimumab 40 mg Eow vs DB Placebo ew; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Chi-squared

2. Primary Outcome: Change From Baseline in Modified Total Sharp X-ray Score at Week 52
Description: Modified total Sharp x-ray score (mTSS) is a measure of change in joint health. Radiographs of hands/wrists and feet were obtained at screening and Week 52. Digitized images of these were scored in a blinded manner. Joints were scored for erosions from 0 (no damage) to 5 and for joint space narrowing from 0 (no damage) to 4; scores were added to obtain the mTSS (range = 0 [normal] to 398 [maximal disease]). Large positive change indicates disease progression; small positive/no change indicates slowing/halting of disease progression; and negative change may indicate improvement of disease.
Time Frame: Baseline and Week 52
Population: Full analysis set, defined as all subjects who were randomized and received at least one injection of study drug. Missing values were imputed via linear extrapolation from baseline using data collected at baseline and Week 24 or early termination.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DB Adalimumab 20 mg ew | DB Adalimumab 40 mg Eow | DB Placebo ew
Number analyzed (Participants) | 196 | 183 | 172
Units on a scale | 0.8 (4.9) [-14.5 to 50.5] | 0.1 (4.8) [-37.0 to 23.5] | 2.7 (6.8) [-25.0 to 39.0]
Statistical Analysis 1: Comparison: DB Adalimumab 20 mg ew vs DB Placebo ew; The 3 primary efficacy variables were considered in a hierarchical order, with the change in modified total Sharp x-ray score at Week 52 tested second. Normality was evaluated by applying the Shapiro-Wilk test procedure to the residuals from the parametric model. The final analysis was performed following a non-parametric approach, ranking the results prior to fitting the model; Test type: Superiority or Other; p < 0.001, ANCOVA — An ANCOVA model with baseline erosion scores as the covariate was performed. An overall significance test at alpha =0.05 was done. Pairwise comparisons, each at alpha =0.05 (2-sided), were performed if the overall test was significant
Statistical Analysis 2: Comparison: DB Adalimumab 40 mg Eow vs DB Placebo ew; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]

3. Secondary Outcome: Number of Participants Meeting ACR20 Response Criteria at Week 52
Description: as for outcome 1
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | DB Adalimumab 20 mg ew | DB Adalimumab 40 mg Eow | DB Placebo ew
Number analyzed (Participants) | 212 | 207 | 200
Participants | 116 | 122 | 48
Statistical Analysis 1: Comparison: DB Adalimumab 20 mg ew vs DB Placebo ew; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: DB Adalimumab 40 mg Eow vs DB Placebo ew; Test type: Superiority or Other; p < 0.001, Chi-squared

4. Secondary Outcome: Change From Baseline in Modified Total Sharp X-ray Score at Week 24
Description: Modified total Sharp x-ray score (mTSS) is a measure of change in joint health. Radiographs of hands/wrists and feet were obtained at screening and Week 24. Digitized images of these were scored in a blinded manner. Joints were scored for erosions from 0 (no damage) to 5 and for joint space narrowing from 0 (no damage) to 4; scores were added to obtain the mTSS (range = 0 [normal] to 398 [maximal disease]). Large positive change indicates disease progression; small positive/no change indicates slowing/halting of disease progression; and negative change may indicate improvement of disease.
Time Frame: Baseline and Week 24
Population: Full analysis set, defined as all subjects who were randomized and received at least one injection of study drug. Missing values were imputed via linear extrapolation from baseline using data collected at baseline and Week 52.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DB Adalimumab 20 mg ew | DB Adalimumab 40 mg Eow | DB Placebo ew
Number analyzed (Participants) | 196 | 183 | 172
Units on a scale | 0.6 (4.9) | 0.3 (4.5) | 1.3 (3.7)
Statistical Analysis 1: Comparison: DB Adalimumab 20 mg ew vs DB Placebo ew; Test type: Superiority or Other; p < 0.01, ANCOVA
Statistical Analysis 2: Comparison: DB Adalimumab 40 mg Eow vs DB Placebo ew; Test type: Superiority or Other; p < 0.001, ANCOVA

5. Secondary Outcome: Change From Baseline in the Disability Index of the Health Assessment Questionnaire (HAQ) at Week 24
Description: Subjects assessed their ability to perform the following tasks: 1) dress/groom; 2) arise; 3) eat; 4) walk; 5) reach; 6) grip; 7) maintain hygiene; and 8) maintain daily activity. Subjects assessed their ability to do these tasks over the past week by marking their response on a questionnaire. Possible responses/scores included the following: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Negative mean changes from baseline in the disability index of the HAQ indicated improvement.
Time Frame: Baseline and Week 24
Population: Full analysis set, defined as all subjects who were randomized and received at least one injection of study drug. LOCF data analysis was used for missing values.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DB Adalimumab 20 mg ew | DB Adalimumab 40 mg Eow | DB Placebo ew
Number analyzed (Participants) | 212 | 204 | 198
Units on a scale | -0.60 (0.53) | -0.56 (0.52) | -0.24 (0.52)
Statistical Analysis 1: Comparison: DB Adalimumab 20 mg ew vs DB Placebo ew; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: DB Adalimumab 40 mg Eow vs DB Placebo ew; Test type: Superiority or Other; p < 0.001, ANCOVA

6. Primary Outcome: Change From Baseline in the Disability Index of the Health Assessment Questionnaire (HAQ) at Week 52
Description: as for outcome 5
Time Frame: Baseline and Week 52
Population: Full analysis set, defined as all subjects who were randomized and received at least one injection of study drug. Last observation carried forward (LOCF) data analysis was used for missing values.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DB Adalimumab 20 mg ew | DB Adalimumab 40 mg Eow | DB Placebo ew
Number analyzed (Participants) | 212 | 204 | 198
Units on a scale | -0.61 (0.55) | -0.59 (0.57) | -0.25 (0.56)
Statistical Analysis 1: Comparison: DB Adalimumab 20 mg ew vs DB Placebo ew; The 3 primary efficacy variables were considered in a hierarchical order, with the change from baseline in the HAQ at Week 52 tested last. The difference among all treatment groups was assessed using ANCOVA with the baseline value as the covariate. If this was significant (p<=0.05), pairwise comparisons between each adalimumab dose group and placebo were evaluated using the same method; Test type: Superiority or Other; p < 0.001, ANCOVA — Normality was evaluated by applying the Shapiro-Wilk test to residuals from the parametric model. The final analysis was performed using a parametric approach
Statistical Analysis 2: Comparison: DB Adalimumab 40 mg Eow vs DB Placebo ew; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 1]

7. Secondary Outcome: Maintenance of the Disability Index of the HAQ at Week 52 for Participants Who Were Responders at Week 12 or Week 24
Description: Subjects assessed their ability to perform the following tasks: 1) dress/groom; 2) arise; 3) eat; 4) walk; 5) reach; 6) grip; 7) maintain hygiene; and 8) maintain daily activity. Subjects assessed their ability to do these tasks over the past week by marking their response on a questionnaire. Possible responses/scores included the following: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Responders had a >= 0.22-unit decrease (improvement) in HAQ scores from baseline to Week 12 or 24.
Time Frame: Week 52
Population: Full analysis set, defined as all subjects who were randomized and received at least one injection of study drug. Subjects who were responders at Week 12 or 24 were evaluated to determine whether the response was maintained. LOCF data analysis was used for missing values.
Measure: Number; unit: Participants
Arm/Group | DB Adalimumab 20 mg ew | DB Adalimumab 40 mg Eow | DB Placebo ew
Number analyzed (Participants) | 212 | 207 | 200
Participants
  Maintained Response | 130 | 121 | 73
  Did Not Maintain Response | 7 | 4 | 9
Statistical Analysis 1: Comparison: DB Adalimumab 20 mg ew vs DB Placebo ew; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: DB Adalimumab 40 mg Eow vs DB Placebo ew; Test type: Superiority or Other; p < 0.001, Chi-squared

8. Secondary Outcome: Maintenance of ACR20 Response at Week 52 for Participants Who Were ACR20 Responders at Week 24
Description: as for outcome 1
Time Frame: Week 52
Population: Full analysis set, defined as all subjects who were randomized and received at least one injection of study drug. Subjects who were ACR20 responders at Week 24 were evaluated to determine whether the response was maintained. Observed data were analyzed.
Measure: Number; unit: Participants
Arm/Group | DB Adalimumab 20 mg ew | DB Adalimumab 40 mg Eow | DB Placebo ew
Number analyzed (Participants) | 129 | 131 | 59
Participants
  Maintained Response | 99 | 111 | 32
  Did Not Maintain Response | 21 | 12 | 23
  Missing | 9 | 8 | 4

9. Secondary Outcome: Number of Participants With a Continuous ACR70 Response for 6 Months During 52 Weeks of Treatment
Description: Patients were responders if they had: >= 70% improvement in tender joint count; >= 70% improvement in swollen joint count; and >= 70% improvement in at least 3 of 5 remaining ACR core measures: patient assessment of pain; patient global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and acute phase reactant: C-reactive protein. Patients withdrawing early or receiving additional disease-modifying anti-rheumatic drugs (DMARDs) after Week 16 were non-responders.
Time Frame: Baseline through Week 52
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | DB Adalimumab 20 mg ew | DB Adalimumab 40 mg Eow | DB Placebo ew
Number analyzed (Participants) | 212 | 207 | 200
Participants | 20 | 18 | 3
Statistical Analysis 1: Comparison: DB Adalimumab 20 mg ew vs DB Placebo ew; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: DB Adalimumab 40 mg Eow vs DB Placebo ew; Test type: Superiority or Other; p < 0.001, Chi-squared

10. Secondary Outcome: Time to First Response According to ACR20 Criteria - Number of Participants Meeting ACR20 Criteria for the First Time at Each Time Point
Description: as for outcome 1
Time Frame: Baseline through Week 52
Population: Full analysis set, defined as all subjects who were randomized and received at least one injection of study drug. Observed data were analyzed. The number of subjects meeting ACR20 response criteria for the first time at each time point is presented.
Measure: Number; unit: Participants
Arm/Group | DB Adalimumab 20 mg ew | DB Adalimumab 40 mg Eow | DB Placebo ew
Number analyzed (Participants) | 212 | 207 | 200
Participants
  Non-responder | 25 | 29 | 81
  Week 2 | 69 | 53 | 26
  Week 4 | 48 | 48 | 30
  Week 8 | 29 | 33 | 21
  Week 12 | 17 | 23 | 14
  Week 16 | 7 | 8 | 12
  Week 20 | 8 | 7 | 3
  Week 24 | 2 | 2 | 7
  Week 32 | 4 | 2 | 2
  Week 40 | 0 | 2 | 1
  Week 48 | 1 | 0 | 2
  Week 52 | 2 | 0 | 1

11. Secondary Outcome: Time to First Response According to ACR50 Criteria - Number of Participants Meeting ACR50 Criteria for the First Time at Each Time Point
Description: Patients were responders if they had: >= 50% improvement in tender joint count; >= 50% improvement in swollen joint count; and >= 50% improvement in at least 3 of 5 remaining ACR core measures: patient assessment of pain; patient global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and acute phase reactant: C-reactive protein. Patients withdrawing early or receiving additional disease-modifying anti-rheumatic drugs (DMARDs) after Week 16 were non-responders.
Time Frame: Baseline through Week 52
Population: Full analysis set, defined as all subjects who were randomized and received at least one injection of study drug. Observed data were analyzed. The number of subjects meeting ACR50 response criteria for the first time at each time point is presented.
Measure: Number; unit: Participants
Arm/Group | DB Adalimumab 20 mg ew | DB Adalimumab 40 mg Eow | DB Placebo ew
Number analyzed (Participants) | 212 | 207 | 200
Participants
  Non-responder | 71 | 69 | 135
  Week 2 | 18 | 13 | 4
  Week 4 | 17 | 26 | 6
  Week 8 | 26 | 25 | 6
  Week 12 | 25 | 21 | 10
  Week 16 | 23 | 21 | 8
  Week 20 | 16 | 10 | 9
  Week 24 | 7 | 7 | 3
  Week 32 | 4 | 7 | 8
  Week 40 | 3 | 2 | 6
  Week 48 | 1 | 3 | 3
  Week 52 | 1 | 3 | 2

12. Secondary Outcome: Time to First Response According to ACR70 Criteria - Number of Participants Meeting ACR70 Criteria for the First Time at Each Time Point
Description: as for outcome 9
Time Frame: Baseline through Week 52
Population: Full analysis set, defined as all subjects who were randomized and received at least one injection of study drug. Observed data were analyzed. The number of subjects meeting ACR70 response criteria for the first time at each time point is presented.
Measure: Number; unit: Participants
Arm/Group | DB Adalimumab 20 mg ew | DB Adalimumab 40 mg Eow | DB Placebo ew
Number analyzed (Participants) | 212 | 207 | 200
Participants
  Non-responder | 126 | 120 | 177
  Week 2 | 5 | 5 | 2
  Week 4 | 5 | 6 | 3
  Week 8 | 11 | 7 | 1
  Week 12 | 14 | 16 | 2
  Week 16 | 15 | 9 | 1
  Week 20 | 9 | 11 | 2
  Week 24 | 4 | 11 | 2
  Week 32 | 9 | 8 | 3
  Week 40 | 4 | 4 | 2
  Week 48 | 4 | 6 | 3
  Week 52 | 6 | 4 | 2

13. Secondary Outcome: Estimated Yearly Progression of Rheumatoid Arthritis
Description: Estimated yearly progression was defined as modified total Sharp x-ray score at baseline divided by duration of rheumatoid arthritis disease at baseline. Actual progression during the study was defined as modified total Sharp x-ray score at Week 52 minus modified total Sharp x-ray score at baseline divided by the duration of the study. The range of scores for the modified total Sharp x-ray score was 0 (normal) to 398 (maximal disease).
Time Frame: Baseline and Week 52
Population: Full analysis set, defined as all subjects who were randomized and received at least one injection of study drug. Missing values were imputed via linear extrapolation from baseline.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DB Adalimumab 20 mg ew | DB Adalimumab 40 mg Eow | DB Placebo ew
Number analyzed (Participants) | 200 | 194 | 184
Units on a scale
  Estimated yearly progression | 11.11 (16.75) | 9.46 (10.42) | 9.97 (12.84)
  Actual progression during study | 0.77 (4.90) | 0.09 (4.75) | 2.66 (6.73)
Statistical Analysis 1: Comparison: DB Adalimumab 20 mg ew vs DB Placebo ew; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: DB Adalimumab 40 mg Eow vs DB Placebo ew; Test type: Superiority or Other; p < 0.001, ANCOVA

14. Other Pre Specified Outcome: Baseline Measure: Gender - Female/Male - for the Any Adalimumab Through Year 10 Group (Intent-to-Treat)
Description: Gender (female/male) recorded at Baseline for the Intent-to-Treat population (the Any Adalimumab Through Year 10 group) of the study. This measure was not included in the Baseline Characteristics section due to the difficulty of maintaining correct subject numbers and totals in that section.
Time Frame: Baseline for Intent-to-Treat (Any Adalimumab Through Year 10) Group
Population: Participants in the Any Adalimumab Through Year 10 group are intent-to-treat subjects.
Measure: Number; unit: participants
Groups:
- Any Adalimumab Through Year 10: Subjects received at least 1 dose of adalimumab over the 10-year duration of the study (the intent-to-treat population, N = 553).
Arm/Group | Any Adalimumab Through Year 10
Number analyzed (Participants) | 553
participants
  Female | 413
  Male | 140

15. Other Pre Specified Outcome: Baseline Measure: Age Categories for the Any Adalimumab Through Year 10 Group (Intent-to-Treat)
Description: Age recorded at Baseline, reported by category, for the Intent-to-Treat population (the Any Adalimumab Through Year 10 group) of the study. This measure was not included in the Baseline Characteristics section due to the difficulty of maintaining correct subject numbers and totals in that section.
Time Frame: Baseline for Intent-to-Treat (Any Adalimumab Through Year 10) Group
Population: Participants in the Any Adalimumab Through Year 10 group are intent-to-treat subjects.
Measure: Number; unit: participants
Arm/Group | Any Adalimumab Through Year 10
Number analyzed (Participants) | 553
participants
  < 40 years | 50
  Between 40 and 64 years | 361
  Between 65 and 74 years | 117
  >= 75 years | 25

16. Other Pre Specified Outcome: Number of Participants Meeting American College of Rheumatology 20% (ACR20) Response Criteria at Week 260
Description: Patients were responders if they had: >= 20% improvement in tender joint count; >= 20% improvement in swollen joint count; and >= 20% improvement in at least 3 of 5 remaining ACR core measures: patient assessment of pain; patient global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and acute phase reactant: C-reactive protein.
Time Frame: Week 260
Population: Participants analyzed were intent-to-treat subjects with non-missing response who remained in the study. All analyses were performed as observed (without imputation).
Measure: Number; unit: Participants
Arm/Group | Any Adalimumab Through Year 10
Number analyzed (Participants) | 290
Participants | 200

17. Other Pre Specified Outcome: Number of Participants Meeting the American College of Rheumatology 20% (ACR20) Response Criteria at Week 520
Description: as for outcome 16
Time Frame: Week 520
Population: Participants analyzed were intent-to-treat subjects with non-missing response who remained in the study. All analyses were performed using data as observed (without imputation).
Measure: Number; unit: participants
Arm/Group | Any Adalimumab Through Year 10
Number analyzed (Participants) | 148
participants | 115

18. Other Pre Specified Outcome: Number of Participants Meeting American College of Rheumatology 50% (ACR50) Response Criteria at Week 260
Description: Patients were responders if they had: >= 50% improvement in tender joint count; >= 50% improvement in swollen joint count; and >= 50% improvement in at least 3 of 5 remaining ACR core measures: patient assessment of pain; patient global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and acute phase reactant: C-reactive protein.
Time Frame: Week 260
Population: Participants analyzed were intent-to-treat subjects with non-missing response who remained in the study. All analyses were performed using data as observed (no imputation).
Measure: Number; unit: participants
Arm/Group | Any Adalimumab Through Year 10
Number analyzed (Participants) | 290
participants | 153

19. Other Pre Specified Outcome: Number of Participants Meeting the American College of Rheumatology 50% (ACR50) Response Criteria at Week 520
Description: as for outcome 18
Time Frame: Week 520
Population: as for outcome 18
Measure: Number; unit: participants
Arm/Group | Any Adalimumab Through Year 10
Number analyzed (Participants) | 148
participants | 100

20. Other Pre Specified Outcome: Number of Participants Meeting the American College of Rheumatology 70% (ACR70) Response Criteria at Week 260
Description: Patients were responders if they had: >= 70% improvement in tender joint count; >= 70% improvement in swollen joint count; and >= 70% improvement in at least 3 of 5 remaining ACR core measures: patient assessment of pain; patient global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and acute phase reactant: C-reactive protein.
Time Frame: Week 260
Population: as for outcome 18
Measure: Number; unit: participants
Arm/Group | Any Adalimumab Through Year 10
Number analyzed (Participants) | 290
participants | 87

21. Other Pre Specified Outcome: Number of Participants Meeting the American College of Rheumatology 70% (ACR70) Response Criteria at Week 520
Description: as for outcome 20
Time Frame: Week 520
Population: as for outcome 18
Measure: Number; unit: participants
Arm/Group | Any Adalimumab Through Year 10
Number analyzed (Participants) | 148
participants | 78

22. Other Pre Specified Outcome: Number of Participants With a Continuous American College of Rheumatology 70% (ACR70) Response for at Least 6 Months Through Year 10
Description: Patients were responders if they had: >=70% improvement in tender joint count; >=70% improvement in swollen joint count; and >=70% improvement in at least 3 of 5 remaining ACR core measures: patient assessment of pain; patient global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and acute phase reactant: C-reactive protein.
Time Frame: Baseline through Week 520
Population: Participants analyzed were intent-to-treat subjects with non-missing response. Analyses were performed using data as observed (no imputation).
Measure: Number; unit: participants
Arm/Group | Any Adalimumab Through Year 10
Number analyzed (Participants) | 535
participants | 159

23. Other Pre Specified Outcome: Number of Participants With at Least a 0.22 Reduction From Baseline in the Health Assessment Questionnaire (HAQ) Disability Index at Week 260
Description: The Health Assessment Questionnaire (HAQ) Disability Index is a self-reported measure of disability, which assesses the patient's ability to perform the following tasks: dress and groom; arise; eat; walk; reach; grip; maintain hygiene; and maintain daily activity. Possible responses/scores are 0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty), and 3 (unable to do). Negative mean changes from Baseline indicate improvement. An improvement of 0.22 in score (a -0.22 or greater reduction from Baseline score) is a minimally clinically significant change.
Time Frame: Week 260
Population: Participants analyzed were intent-to-treat with non-missing response who remained in the study. Baseline was the last non-missing value prior to the first injection of adalimumab. Analyses were performed using data as observed (no imputation).
Measure: Number; unit: participants
Arm/Group | Any Adalimumab Through Year 10
Number analyzed (Participants) | 300
participants | 205

24. Other Pre Specified Outcome: Number of Participants With at Least a 0.22 Reduction From Baseline in the Health Assessment Questionnaire (HAQ) Disability Index at Week 520
Description: as for outcome 23
Time Frame: Week 520
Population: Participants analyzed were intent-to-treat subjects with non-missing response who remained in the study. Baseline was the last non-missing value prior to the first injection of adalimumab. Analyses were performed using data as observed (no imputation).
Measure: Number; unit: participants
Arm/Group | Any Adalimumab Through Year 10
Number analyzed (Participants) | 149
participants | 110

25. Other Pre Specified Outcome: Change From Baseline in the Disability Index of the Health Assessment Questionnaire (HAQ) at Week 260
Description: Subjects assessed their ability to perform the following tasks: 1) dress/groom; 2) arise; 3)eat; 4) walk; 5) reach; 6) grip; 7) maintain hygiene; and 8) maintain daily activity. Subjects assessed their ability to do these tasks over the past week by marking their response on a questionnaire. Possible responses/scores were: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Negative mean changes from Baseline in the disability index of the HAQ indicated improvement.
Time Frame: Baseline and Week 260
Population: Participants analyzed were intent-to-treat subjects with non-missing change who remained in the study. Baseline was the last non-missing value prior to the first injection of adalimumab. Analyses were performed using data as observed (no imputation).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Any Adalimumab Through Year 10
Number analyzed (Participants) | 300
units on a scale | -0.56 (0.62)

26. Other Pre Specified Outcome: Change From Baseline in the Disability Index of the Health Assessment Questionnaire (HAQ) at Week 520
Description: as for outcome 25
Time Frame: Baseline and Week 520
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Any Adalimumab Through Year 10
Number analyzed (Participants) | 149
units on a scale | -0.62 (0.60)

27. Other Pre Specified Outcome: Change From Baseline in Modified Total Sharp X-ray Score at Week 416
Description: Modified total Sharp x-ray score (mTSS) is a measure of change in joint health. Radiographs of hands/wrists and feet were obtained at screening and Week 416. Digitized images of these were scored in a blinded manner. Joints were scored for erosions from 0 (no damage) to 5 and for joint space narrowing from 0 (no damage) to 4; scores were added to obtain the mTSS (range = 0 [normal] to 398 [maximal disease]). Large positive change indicates disease progression; small positive/no change indicates slowing/halting of disease progression; and negative change may indicate improvement of disease.
Time Frame: Baseline and Week 416
Population: Participants in each of the three groups were randomized subjects with non-missing radiographs who remained in the study. Baseline was defined as the value at the first visit. Analyses were performed using data as observed (no imputation).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- DB Adalimumab 20 mg ew/OL Adalimumab 40 mg Eow: Subjects received adalimumab 20 mg every week (ew) during the double-blind (DB) phase, followed by adalimumab every other week (eow) during the open-label (OL) extension, along with concomitant methotrexate (MTX).
- DB Adalimumab 40 mg Eow/OL Adalimumab 40 mg Eow: Subjects received adalimumab 40 mg every other week (eow) during the double-blind (DB) phase, followed by adalimumab 40 mg eow during the open-label (OL) extension phase, along with concomitant methotrexate (MTX).
- DB Placebo ew/OL Adalimumab 40 mg Eow: Subjects received placebo every week (ew) during the double-blind (DB) phase, followed by adalimumab 40 mg every other week (eow) during the open-label (OL) extension phase, along with concomitant methotrexate (MTX).
Arm/Group | DB Adalimumab 20 mg ew/OL Adalimumab 40 mg Eow | DB Adalimumab 40 mg Eow/OL Adalimumab 40 mg Eow | DB Placebo ew/OL Adalimumab 40 mg Eow
Number analyzed (Participants) | 70 | 81 | 53
units on a scale | 1.16 (7.969) | 0.14 (9.310) | 4.83 (10.012)

28. Other Pre Specified Outcome: Change From Baseline in Modified Total Sharp X-ray Score at Week 520
Description: Modified total Sharp x-ray score (mTSS) is a measure of change in joint health. Radiographs of hands/wrists and feet were obtained at screening and Week 520. Digitized images of these were scored in a blinded manner. Joints were scored for erosions from 0 (no damage) to 5 and for joint space narrowing from 0 (no damage) to 4; scores were added to obtain the mTSS (range = 0 [normal] to 398 [maximal disease]). Large positive change indicates disease progression; small positive/no change indicates slowing/halting of disease progression; and negative change may indicate improvement of disease.
Time Frame: Baseline and Week 520
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DB Adalimumab 20 mg ew/OL Adalimumab 40 mg Eow | DB Adalimumab 40 mg Eow/OL Adalimumab 40 mg Eow | DB Placebo ew/OL Adalimumab 40 mg Eow
Number analyzed (Participants) | 70 | 79 | 54
units on a scale | 2.60 (8.822) | 0.72 (10.430) | 6.18 (12.071)

ADVERSE EVENTS:
Time Frame: For the double-blind (DB) phase: Week 0 to Week 52; for the Any Adalimumab Through Year 10 (intent-to-treat [ITT]) group: first adalimumab injection to the last day in Year 10 (for each subject, the day of the last adalimumab injection plus 70 days)
Description: The protocol specified that adverse events (AEs) be summarized by HARTS body system/preferred term (used in the clinical study report and primary publication for the DB phase). AE terms for the DB phase were recoded using MedDRA version 12.1 for purposes of this disclosure. AEs for the Any Adalimumab group were coded using MedDRA version 13.1.
Arm/Group | DB Adalimumab 20 mg ew | DB Adalimumab 40 mg Eow | DB Placebo ew | Any Adalimumab Through Year 10
Serious Adverse Events (participants affected / at risk) | 34/212 | 27/207 | 20/200 | 271/553
Other Adverse Events (participants affected / at risk) | 167/212 | 148/207 | 149/200 | 511/553
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB Adalimumab 20 mg ew (N=212) | DB Adalimumab 40 mg Eow (N=207) | DB Placebo ew (N=200) | Any Adalimumab Through Year 10 (N=553)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 2 | 2
Acute tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 13
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 1 | 7
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 3
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 5
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 6
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 5
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 3
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Chemical poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 4
Cholecystectomy (Surgical and medical procedures) | 1 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 3
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 4
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 2
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 7
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 6
Depression (Psychiatric disorders) | 0 | 0 | 1 | 2
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Escherichia sepsis (Infections and infestations) | 1 | 1 | 0 | 3
Femur fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 6
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 2
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 7
Histoplasmosis (Infections and infestations) | 0 | 1 | 0 | 5
Hysterectomy (Surgical and medical procedures) | 0 | 1 | 0 | 1
Infected skin ulcer (Infections and infestations) | 1 | 0 | 0 | 1
Iodine allergy (Immune system disorders) | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2
Joint dislocation postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 2 | 0 | 0 | 3
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Multiple sclerosis (Nervous system disorders) | 1 | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 10
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 6
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 2
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2
Pelvic mass (General disorders) | 0 | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Pneumonia (Infections and infestations) | 1 | 4 | 1 | 20
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 5
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 5
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Renal vessel disorder (Renal and urinary disorders) | 1 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 35
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0 | 3
Serum sickness (Immune system disorders) | 0 | 0 | 1 | 0
Skin neoplasm excision (Surgical and medical procedures) | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 3
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2
Testicular seminoma (pure) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2
Toe operation (Surgical and medical procedures) | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 3
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 2
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 2
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 2
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 2
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 2
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 1
Mitral valve disease (Cardiac disorders) | 0 | 0 | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 0 | 2
Silent myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2
Cardiac septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Inner ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Enterocele (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric volvulus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrititis (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Gastrointestinal heamorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal infarction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Salivary gland mass (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Cyst rupture (General disorders) | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 0 | 1
Device dislocation (General disorders) | 0 | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 2
Sudden death (General disorders) | 0 | 0 | 0 | 1
Ulcer haemorrhage (General disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 5
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 2
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 3
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Bronchiectasis (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 15
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 1
Enterococal infection (Infections and infestations) | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1
Eye infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 3
Haematoma infection (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster ophthalmic (Infections and infestations) | 0 | 0 | 0 | 1
Histoplasmosis disseminated (Infections and infestations) | 0 | 0 | 0 | 1
Incision site infection (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 1
Liver abscess (Infections and infestations) | 0 | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 7
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1
Meningitis viral (Infections and infestations) | 0 | 0 | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 2
Pneumonia primary atypical (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 5
Sepsis (Infections and infestations) | 0 | 0 | 0 | 4
Sepsis syndrome (Infections and infestations) | 0 | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 2
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 2
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 2
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Back injuury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 4
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin flap necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Hand deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cervix carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 3
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ovarian epithelial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Small intestine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 0 | 2
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 2
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 0 | 4
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 6
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 1
Bladder disorder (Renal and urinary disorders) | 0 | 0 | 0 | 1
Bladder prolapse (Renal and urinary disorders) | 0 | 0 | 0 | 2
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 2
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 2
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 2
Pelvic prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 3
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Rectocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 2
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Ankle operation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Breast prosthesis implantation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Breast reconstruction (Surgical and medical procedures) | 0 | 0 | 0 | 1
Finger amputation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Foot operation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Gastric bypass (Surgical and medical procedures) | 0 | 0 | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 2
Mastectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1
Spinal laminectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1
Angiopathy (Vascular disorders) | 0 | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 3
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 5
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1
Hypertensive emergency (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB Adalimumab 20 mg ew (N=212) | DB Adalimumab 40 mg Eow (N=207) | DB Placebo ew (N=200) | Any Adalimumab Through Year 10 (N=553)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 11 | 15 | 120
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 10 | 9 | 103
Bronchitis (Infections and infestations) | 16 | 7 | 15 | 106
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 16 | 14 | 72
Diarrhoea (Gastrointestinal disorders) | 23 | 20 | 30 | 97
Dizziness (Nervous system disorders) | 11 | 7 | 11 | 63
Influenza (Infections and infestations) | 10 | 6 | 13 | 79
Headache (Nervous system disorders) | 28 | 24 | 10 | 95
Hypertension (Vascular disorders) | 11 | 9 | 4 | 116
Injection site pain (General disorders) | 37 | 37 | 43 | 74
Nausea (Gastrointestinal disorders) | 28 | 19 | 25 | 94
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 11 | 8 | 77
Oedema peripheral (General disorders) | 2 | 11 | 7 | 76
Rash (Skin and subcutaneous tissue disorders) | 12 | 15 | 10 | 83
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 11 | 9 | 42
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 8 | 17 | 51
Upper respiratory tract infection (Infections and infestations) | 35 | 35 | 22 | 225
Urinary tract infection (Infections and infestations) | 16 | 18 | 15 | 118
Vomiting (Gastrointestinal disorders) | 6 | 4 | 12 | 42
Fatigue (General disorders) | 18 | 11 | 15 | 79
Nasopharyngitis (Infections and infestations) | 23 | 24 | 18 | 119
Sinusitis (Infections and infestations) | 21 | 22 | 17 | 150
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 | 8 | 10 | 44
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 10 | 14 | 24 | 123
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 39
Cataract (Eye disorders) | 0 | 0 | 0 | 59
Dry eye (Eye disorders) | 0 | 0 | 0 | 31
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 31
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 40
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 35
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 47
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 51
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 52
Chest pain (General disorders) | 0 | 0 | 0 | 42
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 33
Ear infection (Infections and infestations) | 0 | 0 | 0 | 30
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 35
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 50
Localised infection (Infections and infestations) | 0 | 0 | 0 | 30
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 29
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 32
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 29
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 46
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 35
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 29
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 32
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 38
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 42
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 42
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 48
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 29
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 45
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 45
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 50
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 32
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 32
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 35
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 35
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 29
Depression (Psychiatric disorders) | 0 | 0 | 0 | 71
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 49
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 38
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 28
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection